CLINICAL TRIAL: NCT00488917
Title: Sepsis, Endothelial Function, and Lipids in Critically Ill Patients With Liver Failure (the SELLIFA Study)
Acronym: SELLIFA
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Pierre-François Laterre, MD, Cliniques universitaires Saint-Luc, Université catholique de Louvain
Other Study IDs: SELLIFA-01; B40320072194
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Liver Diseases; Liver Cirrhosis; Sepsis; Critical Illness
Keywords: Liver cirrhosis; acute liver failure; liver transplantation; sepsis, infection; endothelium; lipids; diagnosis; prognosis
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Sepsis; Critical Illness; Liver Failure, Acute; Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, urine, ascites fluid.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to determine the role of new biomarkers in the diagnosis of sepsis in critically-ill patients with liver failure and to correlate the prognosis of these patients with parameters of endothelial function and lipid metabolism.

DETAILED DESCRIPTION:
Early diagnosis of sepsis may be difficult in patients with severe liver failure in the absence of usual warning clinical signs. Furthermore, routine laboratory tests like blood leucocyte count and serum c-reactive protein may be misleading in most of these patients. A great interest is taken in the identification of sepsis biomarkers or sepsis-induced alterations in the inflammation cascade, whose expression is independent of liver function. Determination of such a biomarker may be a useful tool for the early diagnosis of sepsis and may have a prognostic significance in patients with liver failure.

Septic complications in patients with liver failure may induce a disruption of liver microcirculation, which is regulated by several factors acting on endothelial and liver stellate cells. Furthermore, generation of reactive oxygen species results in an oxidative stress on lipids, proteins, and DNA. Lipid peroxidation may contribute to further hepatocellular injury and activation of systemic inflammation cascade. Both endothelial dysfunction and alterations in lipid metabolism may have a role in the prognosis of liver disease and its complications.

The purpose of this prospective observational study is to determine the role of new biomarkers in the diagnosis of sepsis in critically-ill patients with liver failure and to correlate the prognosis of these patients with parameters of endothelial function and lipid metabolism. In addition, the porto-systemic gradient of these parameters will be determined in patients planned for a transjugular intra-hepatic porto-systemic shunt (TIPSS).

An overall number of 120 patients will be enrolled. According to the mode of presentation, the planned number of patients in the different study groups will be as follow : 70 patients with chronic liver failure and acute on chronic liver failure; 20 patients with acute liver failure ; 30 patients post-liver transplantation.

ELIGIBILITY:
Inclusion Criteria :

* All consecutive patients with a diagnosis of chronic liver failure, acute on chronic liver failure, acute liver failure, or post-liver transplantation ;
* Adult patient aged 18 years or above, and less than 85 ;
* Admission to the ICU for an expected period of > 24 hours or elective admission for TIPSS placement ;
* Informed consent of the patient or nearest relative.

Exclusion Criteria :

* Age less than 18 years and more than 85 ;
* Pregnancy, including HELLP syndrome ;
* Active malignancy with metastases (localised hepatocellular carcinoma is not an exclusion criteria);
* Systemic chemotherapy in the last 4 weeks (trans-arterial chemo-embolisation for localised hepatocellular carcinoma is not an exclusion criteria) ;
* Acquired immunodeficiency syndrome and antiretroviral therapy ;
* Refusal of the patient or nearest relative.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care unit
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, MD, Study Director — Cliniques Universitaires St Luc, Université Catholique de Louvain; Yvan Fleury, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires St Luc, Université Catholique de Louvain, Brussels, Belgium